CLINICAL TRIAL: NCT06196710
Title: The Use of Over-the-scope-clips in Large Bleeding Gastro-duodenal Ulcers; a Randomized Comparison to Standard Endoscopic Hemostatic Methods
Brief Title: The Use of OTSC in LBGDU to Standard Endoscopic Hemostatic Methods
Acronym: OTSC-LBGDU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not funded for the project.
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other); West China Hospital (Other); Beijing Friendship Hospital (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, MD, PROFESSOR, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTSC-LBGDU
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Bleeding Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Intervention Model Description: Patients are randomized in a 1:1 ratio to receive; endoscopic treatment using OTSC or standard therapies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Over-the-scope Clips (Experimental): Endoscopic Application of Over-the-scope Clips
  Interventions: Device: Over-the-scope Clips
- standard treatment (Active Comparator): standard treatment of either hemo-clipping or thermo-coagulation with or without pre injection with diluted epinephrine <=20 clips or pulse
  Interventions: Device: Hemo-clipping

INTERVENTIONS:
Device: Over-the-scope Clips — Over-the-scope Clips is mounted onto a transparent cap, which is attached to the tip of the endoscope. To deploy the claw device, a cogwheel at the scope head is turned pulling a trip string. This in turn retracts the cap releasing the OTSC onto the vessels.
  Other Names: OTSC
  Arms: Over-the-scope Clips
Device: Hemo-clipping — Contact thermocoagulation using a 3.3mm probe, hemo-clips, or both. The use of the bipolar device involves firm mechanical compression and coagulation for about 8 seconds.
  Other Names: quick clips; thermo-coagulation
  Arms: standard treatment

SUMMARY:
In managing bleeding gastroduodenal ulcers, endoscopic control of bleeding is the first line treatment-further bleeding after endoscopic hemostasis is associated with a 3-fold increase in mortality. Large ulcer size (> 20 mm) predicts further bleeding. These ulcers erode into arteries of significant size (>2 mm) from either the gastro-duodenal or left gastric arterial complexes. An over-the-scope clip is an endoscopic clamp device with a high tensile strength. It can compress sizeable arteries, and firmly anchor onto the ulcer base avoiding recurrent bleeding from clip dislodgement. It therefore offers secure and durable hemostasis.

In the proposed randomized controlled trial, the investigators hypothesize that after initial endoscopic control of bleeding from large gastro-duodenal ulcers (20 mm in size or more), adding an OTSC can prevent recurrent bleeding and improve patients' outcomes. Investigators enroll patients with bleeding from large ulcers as defined. After initial endoscopic control of bleeding using injection with diluted epinephrine, these patients are randomized, during endoscopy, to receive standard treatment (thermo-coagulation or hemo-clips) or an added OTSC. The primary endpoint is recurrent bleeding over 30 days confirmed on endoscopy. Secondary endpoints include the need for rescue treatment; endoscopic, angiographic embolization or surgery, red blood cell (RBC) transfusion, hospitalization, and bleeding related and all-cause mortality.

DETAILED DESCRIPTION:
Endoscopic hemostatic treatment is the cornerstone of the management of patients with acute nonvariceal upper gastrointestinal bleeding. The current standard in endoscopic hemostasis includes the use of hemo-clips or contact thermal devices with or without pre-injection with diluted epinephrine. However, the failure rate with either method approaches 10%. Further bleeding after endoscopic treatment is associated with a 3-fold increase in mortality. The United Kingdom audit reported a 30% mortality in those who required surgery after failed endoscopic treatment.

Over-the-scope clips (OTSCs) are memory-shaped nitinol clips that are cap-mounted onto the end of an endoscope. They were designed for endoscopic closure of full-thickness mucosal defects. They are being increasingly used for the purpose of hemostasis. When deployed, the OTSC provides firm compression on bleeding vessels of significant sizes (>2mm). The retention rate with OTSCs is high avoiding recurrent bleeding from clip dislodgement.

The OTSCs were first evaluated as a rescue treatment in the German Multicenter Trial (Stop the Bleeding or STING 1 trial). The trial enrolled patients with bleeding from their ulcers refractory to standard endoscopic treatment and randomized them to receive either OTSC or further treatment with standard methods. Further bleeding within 30 days after either treatment was 15.2% and 57.6% respectively.

The primary use of OTSC i.e. as the first hemostatic device has been studied in several trials. (see Table 1).

Table 1: Further bleeding in 30 days Author, Year OTSC Standard Treatment

Jensen 2021 1 /25, 4% 8/ 28, 28.6%

Meier 2022 4/ 44, 8.3% 14/ 52, 26.9%

Chan 2023 (ulcers 15 mm or more) 5/ 50, 10% 9/ 50, 18%

Lau 2023 3/ 93, 3.2% 14/ 97, 14.6%

All of the above studies except one showed significant differences in the rate of further bleeds within 30 days in favor of the use of OTSC.

The role of OTSCs in larger gastroduodenal ulcers remains inconclusive. Chan studied exclusively ulcers of 15 mm or above in size. In this study, the use of OTSC did not significantly reduce further bleeds compared to standard treatment (rate of further bleeding 10% vs. 18%). There may have been two reasons to explain a negative trial; first, there were 4 primary failures with the use of OTSC (4/ 50, 8%). Two OTSCs did not fully encompass the vessels. In 2 cases, there were persistent bleeds despite the placement of OTSCs. The authors attributed the failure with the use of OTSC to a learning curve issue. Recurrent bleeds occurred in 2 of 46 (4.4%) after OTSC and 9 of 48 (18.8%) after standard treatments. Because of a small sample size and likely a type 2 error, the overall difference did not reach statistical significance. Gastroduodenal ulcers of 20 mm or more in size are the most critical predictor of further bleeds and failures with endoscopic treatment. These ulcers erode into major arterial complexes to the gastroduodenal and left gastric arteries. An OTSC appears to work well in such ulcers. In a post hoc analysis of our randomized controlled trial (RCT) on the primary use of OTSCs, further bleeds among ulcers 20 mm or larger occurred in 1 of 10 after OTSC treatment compared to 5 of 9 after standard treatment. Because of the inconclusive and conflicting results from the above trials regarding the efficacy of OTSC in high-risk (20mm or larger in size) bleeding gastroduodenal ulcers, investigators propose a randomized controlled trial with the hypothesis that OTSC is superior to standard treatment in bleeding gastroduodenal ulcers 20mm or greater in size. Investigators argue that OTSC should be the primary treatment of choice for ulcers of such size.

Research methods Trial Design and Organisation This study is an investigator-initiated multicentre trial. The participating centers are tertiary referral university hospitals with a high case volume. These include the Prince of Wales Hospital, Hua-Xi Hospital of Szechuan University, Beijing Friendship Hospital, the first affiliated Hospital of Nanchang University, Nanfang Hospital from China, and the King Chulalongkorn Memorial Hospital in Thailand. These hospitals have substantial experience with the use of OTSC and participated in earlier and ongoing clinical trials that evaluate the use of OTSC.

Investigators will obtain approval from the institutional review board in each participating hospital.

The joint Chinese University of Hong Kong-New Territories East Cluster Clinical Research Ethics Committee oversees the trial execution. Senior physicians from the committee adjudicate outcomes and review serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted with acute upper gastrointestinal bleeding (melena, hematemesis, or decrease in hemoglobin level with or without hypotension).
* large gastro-duodenal ulcers (20 mm in size or more)
* active bleeding (pulsatile or Forrest Ia bleeding, oozing from a visible vessel, or Forrest Ib bleeding) or a nonbleeding visible vessel (Forrest IIa lesion). Clots overlying bleeding lesions are injected with diluted epinephrine and then irrigated or elevated using a cheese-wiring technique. If a vessel is then unveiled, we can proceed with randomization.

Exclusion Criteria:

* patients with esophagogastric varices
* pregnant or lactating women
* patients who cannot provide written consent
* moribund from their co-morbid illnesses and are not considered for active treatment.

Ages: 18 Years to 111 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
bleeding free probability in 30 days after randomization | 30 days
  further bleeding defined by the composite of failure to control bleeding after assigned endoscopic treatment and recurrent bleeding.

SECONDARY OUTCOMES:
failure to control bleeding with assigned endoscopic treatment and recurrent bleeding after initial hemostasis | 30 days
  failure to control bleeding during the first endoscopy was defined as persistent or active bleeding after the attempted application of assigned endoscopic treatment. Recurrent bleeding was defined by fresh hematemesis, fresh melena, or hematochezia with hemodynamic instability (systolic blood pressure <90 mm Hg, heart rate >110 beats/min), and/or decrease in hemoglobin level greater than 20 g/L in 24 hours after transfusion to around 80 g/L. Patients who fulfill the clinical criteria of recurrent bleeding undergo urgent endoscopy. Recurrent bleeding requires endoscopic confirmation showing fresh blood in the gastroduodenal tract and active bleeding from a previously treated ulcer.
number of participants using angiographic treatment | 30 days
  angiogram with embolization to bleeding vessel if primary failure or rebleeding
number of participants using surgical treatment | 30 days
  surgical treatment if primary failure or rebleeding
second endoscopic attempts at hemostasis | 30 days
  attempts at hemostasis if primary failure or rebleeding.

OTHER OUTCOMES:
red cell transfusion | 30 days
  amount of total blood transfusion
number of days in the hospital | 30 days
  hospital stay
number of days in intensive care unit (ICU) | 30 days
  ICU stay
rate of bleeding-related or all-cause deaths | 30 days
  bleeding-related or all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: YUN WONG LAU, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barkun AN, Almadi M, Kuipers EJ, Laine L, Sung J, Tse F, Leontiadis GI, Abraham NS, Calvet X, Chan FKL, Douketis J, Enns R, Gralnek IM, Jairath V, Jensen D, Lau J, Lip GYH, Loffroy R, Maluf-Filho F, Meltzer AC, Reddy N, Saltzman JR, Marshall JK, Bardou M. Management of Nonvariceal Upper Gastrointestinal Bleeding: Guideline Recommendations From the International Consensus Group. Ann Intern Med. 2019 Dec 3;171(11):805-822. doi: 10.7326/M19-1795. Epub 2019 Oct 22. PMID 31634917
- [Background] Hearnshaw SA, Logan RF, Lowe D, Travis SP, Murphy MF, Palmer KR. Acute upper gastrointestinal bleeding in the UK: patient characteristics, diagnoses and outcomes in the 2007 UK audit. Gut. 2011 Oct;60(10):1327-35. doi: 10.1136/gut.2010.228437. Epub 2011 Apr 13. PMID 21490373
- [Background] Schmidt A, Golder S, Goetz M, Meining A, Lau J, von Delius S, Escher M, Hoffmann A, Wiest R, Messmann H, Kratt T, Walter B, Bettinger D, Caca K. Over-the-Scope Clips Are More Effective Than Standard Endoscopic Therapy for Patients With Recurrent Bleeding of Peptic Ulcers. Gastroenterology. 2018 Sep;155(3):674-686.e6. doi: 10.1053/j.gastro.2018.05.037. Epub 2018 May 24. PMID 29803838
- [Background] Jensen DM, Kovacs T, Ghassemi KA, Kaneshiro M, Gornbein J. Randomized Controlled Trial of Over-the-Scope Clip as Initial Treatment of Severe Nonvariceal Upper Gastrointestinal Bleeding. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2315-2323.e2. doi: 10.1016/j.cgh.2020.08.046. Epub 2020 Aug 20. PMID 32828873
- [Background] Meier B, Wannhoff A, Denzer U, Stathopoulos P, Schumacher B, Albers D, Hoffmeister A, Feisthammel J, Walter B, Meining A, Wedi E, Zachaus M, Pickartz T, Kullmer A, Schmidt A, Caca K. Over-the-scope-clips versus standard treatment in high-risk patients with acute non-variceal upper gastrointestinal bleeding: a randomised controlled trial (STING-2). Gut. 2022 Jul;71(7):1251-1258. doi: 10.1136/gutjnl-2021-325300. Epub 2022 Mar 23. PMID 35321938
- [Background] Lau JYW, Li R, Tan CH, Sun XJ, Song HJ, Li L, Ji F, Wang BJ, Shi DT, Leung WK, Hartley I, Moss A, Yu KYY, Suen BY, Li P, Chan FKL. Comparison of Over-the-Scope Clips to Standard Endoscopic Treatment as the Initial Treatment in Patients With Bleeding From a Nonvariceal Upper Gastrointestinal Cause : A Randomized Controlled Trial. Ann Intern Med. 2023 Apr;176(4):455-462. doi: 10.7326/M22-1783. Epub 2023 Mar 7. PMID 36877964
- [Background] Chan S, Pittayanon R, Wang HP, Chen JH, Teoh AY, Kuo YT, Tang RS, Yip HC, Ng SKK, Wong S, Mak JWY, Chan H, Lau L, Lui RN, Wong M, Rerknimitr R, Ng EK, Chiu PWY. Use of over-the-scope clip (OTSC) versus standard therapy for the prevention of rebleeding in large peptic ulcers (size >/=1.5 cm): an open-labelled, multicentre international randomised controlled trial. Gut. 2023 Apr;72(4):638-643. doi: 10.1136/gutjnl-2022-327007. Epub 2022 Oct 28. PMID 36307177
- [Background] Elmunzer BJ, Young SD, Inadomi JM, Schoenfeld P, Laine L. Systematic review of the predictors of recurrent hemorrhage after endoscopic hemostatic therapy for bleeding peptic ulcers. Am J Gastroenterol. 2008 Oct;103(10):2625-32; quiz 2633. doi: 10.1111/j.1572-0241.2008.02070.x. Epub 2008 Aug 5. PMID 18684171
- [Background] Vergara M, Bennett C, Calvet X, Gisbert JP. Epinephrine injection versus epinephrine injection and a second endoscopic method in high-risk bleeding ulcers. Cochrane Database Syst Rev. 2014 Oct 13;2014(10):CD005584. doi: 10.1002/14651858.CD005584.pub3. PMID 25308912
- [Background] Lau JYW, Pittayanon R, Wong KT, Pinjaroen N, Chiu PWY, Rerknimitr R, Holster IL, Kuipers EJ, Wu KC, Au KWL, Chan FKL, Sung JJY. Prophylactic angiographic embolisation after endoscopic control of bleeding to high-risk peptic ulcers: a randomised controlled trial. Gut. 2019 May;68(5):796-803. doi: 10.1136/gutjnl-2018-316074. Epub 2018 May 25. PMID 29802172
- [Background] Casagrande JT, Pike MC. An improved approximate formula for calculating sample sizes for comparing two binomial distributions. Biometrics. 1978 Sep;34(3):483-6. No abstract available. PMID 719125